CLINICAL TRIAL: NCT01101269
Title: Effect of Angiotensin Converting Enzyme Inhibitor, Lisinopril, on Renal Blood Flow and Its Correlation With Proteinuria Reduction in Subjects With Type 2 Diabetes and Kidney Disease (KXK005).
Brief Title: Effect of Angiotensin Converting Enzyme Inhibitor, Lisinopril, on Renal Blood Flow and Its Correlation With Proteinuria Reduction in Subjects With Type 2 Diabetes and Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Kambiz Kalantarinia, MD, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14815
Record Dates: First submitted 2010-04-06; First posted 2010-04-09 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
Keywords: Diabetic nephropathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies | interventions — Angiotensin-Converting Enzyme Inhibitors; Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with diabetic nephropathy (Experimental): Renal blood flow (RBF) will be measured using contrast enhanced ultrasound (CEU) and urine protein will be measured both on and off angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB).
  Interventions: Drug: ACEI or ARB
- Healthy volunteers (Active Comparator): Renal blood flow (RBF) will be measured using contrast enhanced ultrasound (CEU) and urine protein will be measured both on and off angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB).
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: ACEI or ARB — Subjects will be asked to discontinue their usual ACE inhibitor or Angiotensin Receptor Blocker (ARB) for ten days, undergo a CEU using Definity (for renal blood flow assessment) as the contrast agent, then resume their usual ACEI or ARB for ten days, then undergo another CEU using Definity as the contrast agent.
  Arms: Subjects with diabetic nephropathy
Drug: Lisinopril — Subjects will be undergo a CEU using Definity (for renal blood flow assessment) as the contrast agent, then take Lisinopril 10 mg every day for 7 days, after which they will undergo another CEU using Definity as the contrast agent.
  Arms: Healthy volunteers

SUMMARY:
The purpose of the study is to investigate the effect of a blood pressure medication, Lisinopril, or similar drugs in that class, on the flow of blood to the kidneys. In this study, we will compare blood flow to the kidneys in healthy people that do not have diabetes or kidney disease with people that have diabetes and evidence of kidney disease.

DETAILED DESCRIPTION:
Blockers of renin angiotensin aldosterone system (RAAS) are considered the standard of care in treatment of diabetic nephropathy. Their effects are thought to be through multiple mechanisms, including reducing intraglomerular pressure. However, due to the lack of a sensitive, practical and noninvasive method of monitoring renal hemodynamics, the magnitude of hemodynamic effects of these agents and its contribution to proteinuria reduction has not been studied in humans. At the same time, it is not clear if treatment with blockers of the RAAS have similar renal hemodynamic effects in individuals with and without diabetes and kidney disease.

Up to 36 subjects with type 2 diabetes and more than 150 mg of proteinuria who are on stable doses of ACE inhibitors or angiotensin receptor blockers (ARBs) and up to 18 healthy volunteers will be enrolled in this study. Subjects with type 2 diabetes will be asked to stop their ACE inhibitor or ARB medications for 10 days. Between 7 to 10 days after stopping these medications renal blood flow (RBF) will be measured using contrast enhanced ultrasound (CEU) and urine protein will be measured as well for comparison to baseline. Subjects' ACE inhibitors or ARB will be restarted and RBF measurement using CEU and measurement of urine protein excretion will be repeated after 7 days. For comparison, RBF will be measured by CEU in up to 18 healthy volunteers. They will then be started on Lisinopril 10 mg orally once a day for 7 days. On day 7 RBF measurement will be repeated to assess the effect of ACE inhibitors on RBF in healthy individuals as compared to those with diabetic nephropathy.

ELIGIBILITY:
Inclusion For subjects with diabetic nephropathy,

1. Adults (ages 40 - 75 years)
2. Diagnosis of type 2 diabetes for more than 5 years
3. Evidence of diabetic nephropathy as evidenced by

   a. More than 150 mg of proteinuria per day in a 24-hour urine collection, or a spot morning urine protein to creatinine of greater than 0.15, or a spot morning urine albumin to creatinine ratio greater than 100 confirmed on two separate occasions within 12 months
4. Treatment with a blocker of the renin -angiotensin-aldosterone system (either ACE inhibitor or ARB)

For healthy controls,

1. Adults (ages 40 - 75 years)
2. Good general health

Exclusion For subjects with diabetic nephropathy,

1. Type 1 diabetes
2. Glomerular filtration rate less than 40 ml/min/1.73 m2 by MDRD formula
3. Hemoglobin A1C greater than 10%
4. Blood pressure greater than 150/90 mm Hg or less than 100/55 mm Hg
5. History of kidney transplantation
6. Oxygen saturation is less than 80%
7. History of unstable cardiopulmonary conditions, known intracardiac shunts, or pulmonary hypertension
8. History of active cancer within the last 3 years

For healthy controls,

1. History or clinical evidence of any chronic disease
2. Chronic and regular use of any medications except for oral contraceptives and vitamins
3. Clinically significant abnormal screening laboratory values
4. Pregnancy or lactation for women
5. Blood pressure at screening visit less than 110/60
6. History of unstable cardiopulmonary conditions, known intracardiac shunts, or pulmonary hypertension
7. History of active cancer within the last 3 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in renal blood flow (RBF) | Study day 10
  We will use Contrast Enhanced Ultrasound using Definity as the contrast agent to monitor changes in renal blood flow (RBF).
Change in renal blood flow (RBF) | Compared to Study Day 17

SECONDARY OUTCOMES:
Change in Proteinuria | Study day 10
Change in Proteinuria | Compared to study day 17

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Kalantarinia, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States